CLINICAL TRIAL: NCT06153212
Title: Regenerative Treatment of Peri-implantitis: A Comparison of the Reinforced PTFE Mesh (RPM) and the Collagen Membrane in the Submerged Approach: a Randomized Controlled Clinical Trial
Brief Title: Regenerative Treatment of Peri-implantitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Osteogenics Biomedical (Industry)
Responsible Party: Principal Investigator, Muhammad Saleh, Clinical Assistant Professor, Periodontics and Oral Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00169735
Record Dates: First submitted 2023-11-20; First posted 2023-12-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTFE Mesh Membrane (Experimental): A reinforced PTFE Mesh membrane will be used to cover the bone graft.
  Interventions: Procedure: Membrane placement with bone grafting
- Collagen membrane (Active Comparator): A collagen membrane will be used to cover the bone graft.
  Interventions: Procedure: Membrane placement with bone grafting

INTERVENTIONS:
Procedure: Membrane placement with bone grafting — The diseased dental implant will be cleaned and the bone defect will be filled with bone graft and covered by a membrane.

SUMMARY:
The purpose of this study is to study the use of a new type of d-PTFE membrane called reinforced PTFE Mesh (RPM) with dental surgery. The regenerative outcomes of RPM membranes and collagen membrane for surgical reconstructive treatment of peri-implantitis (gum disease around implants) will be compared.

DETAILED DESCRIPTION:
Peri-implantitis is an inflammatory response that leads to irreversible loss of implant supporting bone. This study will investigate the regenerative outcomes obtained with two membranes for surgical reconstructive treatment of peri-implantitis defects when the implant is submerged and primary wound closure is obtained. In one group the newly designed d-PTFE membrane with macropores, known as the RPM membrane will be utilized, which will be compared to the traditional collagen membrane used in the other group. The clinical, radiographic, and histologic outcomes for the regenerative treatment of peri-implantitis when utilizing the same bone graft in combination with either a collagen membrane or the RPM will be evaluated via a parallel-arm randomized controlled clinical trial.

32 patients with peri-implantitis will be recruited and randomized to receive peri-implantitis treatment with either a collagen membrane or an RPM membrane.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Physical status according to the American Society of Anesthesiology (ASA) I or II, which include patients who are systematically healthy or may suffer from mild to moderate, however well-controlled systemic diseases.
* Subjects having at least one dental implant with peri-implantitis according to the definition proposed by the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions (Berglundh et al., 2018):
* Full-mouth plaque score and full-mouth bleeding score ≤ 20% (measured at four sites per tooth)
* Correct 3-dimensional implant positioning, or buccal position ≤ 1 mm
* Implants which have been in function for at least 6 months

Exclusion Criteria:

* A clearly mal-positioned dental implant
* Significant interproximal horizontal bone loss (more than 50% of implant fixture length)
* A mobile dental implant
* Presence of uncontrolled or untreated periodontal disease
* More than 2 weeks usage of antibiotics in the past two months
* Subjects taking medications known to modify bone metabolism or those that can interfere with the normal wound healing (such as bisphosphonates, corticosteroids, hormone replacement therapy, parathyroid hormone, denosumab, strontium ranelate, etc.), or those with uncontrolled systemic diseases or conditions that may similarly affect the patient's healing (osteoporosis, osteopenia, hyperparathyroidism, Paget's disease, uncontrolled diabetes (HBA1c > 8)).
* Pregnant subjects or individuals attempting to get pregnant (self-reported)
* Subjects smoking more than 10 cigarettes a day, or those with a history of drug or alcohol abuse (self-reported)
* Subjects unable to maintain adequate oral hygiene (O'Leary plaque index more than 50%) (O'Leary et al., 1972)
* Any other contraindications for undergoing periodontal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Probing depth measurements in millimeters | About 5 weeks before baseline surgery and at 8.5 months after baseline surgery.
  To compare probing depth measurements using a periodontal probe after peri-implantitis treatment
Bone measurements in millimeters | Baseline and 8 months after baseline surgery
  Bone measurements obtained from CBCT

SECONDARY OUTCOMES:
Clinical attachment levels in millimeters | 8 months after baseline surgery
  To compare clinical attachment measurements using a periodontal probe from baseline to the final follow-up visit
Marginal bone levels in millimeters at the implant site | 8 months after baseline surgery
  To compare marginal bone measurements from periapical radiographs
Volumetric changes of grafted area in cubic millimeters | 8 months after baseline surgery
  To compare volumetric bone measurements of the grafted areas from CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Saleh, BDS, MSD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States